## Investigator initiated study (IIS)

Principal Investigator: Walter Royal, III, MD

Institution and department: University of Maryland School of Medicine

**Department of Neurology** 

Date: July 30, 2014 Amend 1

1. Title of the proposed study: Clinical Biomarkers of Disease Activity and Treatment Response in Patients with CNS Sarcoidosis Treated with H.P. Acthar<sup>®</sup> Gel

## 2. Hypothesis/Hypotheses:

- a. Treatment with H.P. Acthar® Gel will result in the improvement and long-term stabilization of clinical and radiographic abnormalities that occur in patients with CNS sarcoidosis.
- b. Treatment will be also associated with improvement in measures of quality of life.
- c. Specific immunological abnormalities will be observed in patients pre-treatment that will serve a biomarkers of disease activity. These abnormalities will also improve with treatment.
- 3. Rationale for the study: Sarcoidosis is a chronic and frequently progressive systemic disease that affects the central nervous system (CNS) in approximately 5% of patients (Stern et al., 1985). The hallmark of the disease is the development of chronic inflammation with formation of non-caseating granulomas that can involve the brain parenchyma and meninges and appear as contrast-enhancing mass lesions on magnetic resonance imaging (Miller et al., 1988). The granulomas are primarily comprised of proinflammatory T cells (Th1 cells and Th17 cells) and macrophages which accumulate during the early stages of granuloma formation (Agostini et al., 2002; Co et al., 2004). The inflammation that is generated by these cells is modulated by anti-inflammatory responses mediated by Th2 cells and regulatory T (Treg) cells (Agostini et al., 2002; Miyara et al., 2006) that later appear and populate the outer regions of the granuloma. The presence of Treg cells are of particular interest since these cell are also detected in high numbers in peripheral blood and the immune suppression that results may underlie the occurrence of anergy in patients with the disease (Miyara et al., 2006). The treatment of CNS

sarcoidosis involves the use of either corticosteroids or potent immunosuppressive agents, both which can induce severe long-term side effects (Moller, 2003; Stern et al., 2010). The adverse effects of steroids may be avoided by treatment with adrenocorticotropic hormone (ACTH) (Arnason et al., 2013), which is available for patient use as H.P. Acthar® Gel. The efficacy of H.P. Acthar® Gel in the treatment of CNS sarcoidosis and the impact on quality of life have not been previously examined. In addition, little is known regarding the expression of immune markers in CNS sarcoidosis and the association of such markers with disease activity and response to treatment. These issues, therefore, will be explored in the context of this proposal.

## 4. Patient population and estimated sample size:

a. Patients with a diagnosis of CNS sarcoidosis (n=10) will be recruited for these studies.

## 5. Study design:

All patients will be recruited from the inpatient and outpatient services of the University of Maryland School of Medicine Department of Neurology.

## **Criteria for enrollment**

- a. A highly probable diagnosis of sarcoidosis, as determined using the WASOG Sarcoidosis Organ Assessment Instrument (Judson et al., 2014), with involvement limited to the central nervous system.
- b. At the time of enrollment, a history of clinical deterioration based on the development of new symptoms or worsening previously present symptoms with confirmation by clinical examination and objective clinical testing.
- c. If on steroids, on a stable dose of the medication for at least 1 month 3 months.

#### **Assessments**

- a. Administration of questionnaires
  - 1. Patient Determined Disease Steps (PDDS): a disability measurement
  - 2. Montreal Cognitive Assessment (MoCA) and Symbol-Digit Modalities test (SDMT): cognitive assessments
  - 3. Fatigue Assessment Scale (FAS)
  - 4. Short Form-36 Health Survey (SF-36): measures quality of life
  - 5. Work Productivity and Activities Impairment—General Health (WPAI-GH): measures health-related work productivity loss
  - 6. Beck Depression Inventory-II (BDI-II): a depression scale

- b. Brain MRI with and without gadolinium
- c. Phlebotomy
- d. Lumbar puncture

#### **Treatment**

- a. Acthar 80 units subcutaneously per day for 10 days, followed by Acthar 80 units subcutaneously 3 times per week through month 12
- b. Continuation of the patient's previously prescribed CNS sarcoidosis maintenance regimen, as appropriate.
- c. Acthar dose may be adjusted based on the patient's tolerability at the discretion of the investigator.

# <u>Assessments baseline/screening, 4 weeks, 6 months and 12 months post-treatment</u>

- a. Administration of questionnaires
  - i. Patient Determined Disease Steps (PDDS)
  - ii. Montreal Cognitive Assessment (MoCA) and Symbol-Digit Modalities test (SDMT)
  - iii. Fatigue Assessment Scale (FAS)
  - iv. Short Form-36 Health Survey (SF-36)
  - v. Work Productivity and Activities Impairment—General Health (WPAI-GH)
  - vi. Beck Depression Inventory-II (BDI-II)
  - vii. Treatment Satisfaction Questionnaire for Medication (TSQM)
- b. Brain MRI
- c. Phlebotomy

## Assessments at baseline/screening, 3 months and 12 months post-treatment

- a. Lumbar puncture- 3 to 4 teaspoons(15 to 20 ml) of CSF fluid per lumbar puncture
- b. Immunological assessments

#### **Laboratory Assessments**

- a. The following immunological assessments will be performed
  - i. Flow cytometry of mononuclear cells in blood and cerebrospinal fluid (CSF)
  - ii. Activation of peripheral blood mononuclear cells in culture to assess for T cell and monocyte activation responses and for secreted cytokines and chemokines
  - iii. Bio-Plex analysis of levels of secreted cytokines and chemokines in blood, CSF and in cell culture supernatants

### Safety Assessments

| Labs: specific monitoring of serum calcium, potassium, creatinine, cortisol responses and levels, glucose and HbA1c, 1, 25-dihydroxyvitamin D levels Symptoms and signs: specific monitoring for gastrointestinal symptoms (abdominal pain, bloody or black stools, nausea, vomiting or hematemesis), fatigue, edema, hypertension, mood changes, infectious complications |
|---|

# b. Table 1 lists the testing that will be performed on blood (plasma) and CSF samples

| Blood | CSF |
|---|---|
| CBC with differential | Red blood cell count |
| Comprehensive chemistry panel | White blood cell count |
| Angiotensin converting-enzyme level | Protein |
| C-Reactive Protein | Glucose |
| Cortisol (checked 4-24 hours after the Acthar dose) | Angiotensin converting-enzyme level |
| Hemoglobin A1C | IgG index |
| 1, 25-dihydroxyvitamin D | Oligoclonal bands |
| 25-hydroxyvitamin D | Myelin basic protein |
| | Protein electrophoresis |

c. Immune phenotyping of peripheral blood and CSF mononuclear cells, including analysis of Treg cells, and analysis of specific proinflammatory and antiinflammatory subsets by staining for intracytoplasmic cytokine will be performed using flow cytometry as previously described (Royal, III et al., 2009; Royal, III et al., 2007). The cell markers and cytokines for which the cells will be labeled are described in table 2.

| Table 2: Markers for Analyzing Mononuclear Cells by Flow Cytometry | | |
|---|---|---|
| Cell type | Function | Markers |
| T Cells | | |
| 1. CD4+ | | |
| a. Th1 | Proinflammatory | CD3+CD4+Interferon (IFN)-γ |
| b. Th17 | Proinflammatory | CD3+CD4+Interleukin (IL)-17+ |
| c. Th2 | Anti-inflammatory | CD3+CD4+IL-4+ |
| d. Treg | Anti-inflammatory | CD3+CD25+CD127 <sup>Low</sup> |
| 2. CD8+ (cytotoxic) | Proinflammatory | CD3+CD8+ |
| Monocytes (Shi and | | |
| Pamer, 2011) | | |
| 1. Classical | Proinflammatory | CD14++CD16- |
| | (antibacterial) | |
| <ol><li>Intermediate</li></ol> | Proinflammatory (more | CD14+CD16+ |
| | differentiated phenotype) | |
| <ol><li>Non-classical</li></ol> | Proinflammatory (antiviral) | CD14+CD16++ |

d. In vitro activation assays will be performed to assess peripheral blood mononuclear cell proliferative responses and secretion of cytokines, chemokines and other soluble immune factors using approaches that are well established in the lab of the PI (Royal, III et al., 2012), including analyses soluble plasma markers of monocyte activation (Royal W III et al, Clinical and Laboratory Assessments of Monocyte Function and Associations with Cognition and Gender among HIV Infected Individuals in Nigeria, Annual Meeting of the International Society of NeuroVirology, Washington, D.C. October 31, 2013). The cytokines and chemokines are listed in table 3 and will be detected in the University of Maryland Cytokine Core Laboratory by Bio-Plex Assay (Bio-Rad).

| Table 3: Soluble Plasma and CSF Markers | |
|---|---|
| Cell type | Cytokine/Chemokine Marker(s) |
| T Cells (Pan) | IL-2, soluble IL-2 receptor, CXCL8, CCL22 |
| 1. CD4+ | |
| a. Th1 | IFN-γ, IL-12, IL-18 |
| b. Th17 | IL-17 |
| c. Th2 | IL-4, IL-13, IL-10 |
| d. Treg | IL-6, TGF-β |
| 2. CD8+ (cytotoxic) | IFN-γ IL-12, IL-18 |
| Monocytes | TNF-α, IL-1β, IL-10, CCL5, CCL2, CCL-3, CCL4, soluble |
| | CD14, soluble CD16, β2-microblobulin, neopterin, |
| | chitotriosidase |

## 6. Primary end-points:

a. Change in total number of lesions and in the number and size of enhancing lesions 1, 3, 6 months and 12 months relative to baseline

## 7. Secondary end-points:

- a. Change in PDDS, MoCA, SDMT, SF-36, WPAI-GH and BDI-II at 4 weeks, 6 months and 12 months relative to baseline
- b. TSQM scores at 4 weeks and change in TSQM scores at 6 months and 12 months versus baseline

## 8. Exploratory endpoints

a. Change in levels of immune markers at 4 weeks, 6 months and 12 months versus baseline

#### 9. Estimated time line:

- a. Months 0-15: Enrollment and assessment
- **b.** Months 14-18: Initial analysis of clinical laboratory data for presentation at scientific meetings and for publication
- c. Months 18-24: Manuscript preparation and submission

**Schedule of Events (table 4)** 

| Table 4. Schedule of | Screening/ | Follow-up (post treatment initiation) | | | |
|---|---|---|---|---|---|
| Events | Baseline | 1 mo. | 3 mos. | 6 mos. | 12 mos. |
| Informed consent | Х | | | | |
| Medical history | X | | | | |
| Physical exam | X | <u>X</u> | <u>X</u> | <u>X</u> | X |
| Neurological exam | X | <u>X</u> | <u>X</u> | <u>X</u> | X |
| Vital signs | X | Х | Х | Х | Х |
| Clinical laboratory testing | X | <u>X</u> | <u>X</u> | <u>X</u> | X |
| Pregnancy test | X | | | | |
| Inclusion/exclusion criteria | X | | | | |
| MRI | X | Х | Х | Х | Х |
| Phlebotomy | X | Х | Х | Х | Х |
| PDDS | X | Х | Х | Х | Х |
| MoCA/SDMT | X | Х | Х | Х | Х |
| SF-36 | Х | Х | Х | Х | Х |
| WPAI-GH | Х | Х | Х | Х | Х |
| TSQM | Х | Х | Х | Х | Х |
| KPSS | Х | Х | Х | Х | Х |
| Lumbar puncture | Х | | Х | | Х |
| Immune assessments | Х | | Х | | Х |

## 10. Budget (table 5)

| | YR 1 | YR 2 | TOTAL |
|---|---|---|---|
| Clinical laboratory tests (\$250) | 4,500 | 1,500 | 6,000 |
| Pregnancy tests (up to 10 tests; \$18 per test) | 180 | 0 | 180 |
| Other clinical laboratory supplies (250) | 7,500 | 2,500 | 10,000 |
| Lumbar punctures (includes labs) (\$1,200) | 4,500 | 15,000 | 19,500 |
| MRI scans (5 per pt.; 10 pts; \$1,200 per MRI) | 36,000 | 24,000 | 60,000 |
| Immune assays | | | |
| Flow cytometry | 20,000 | 10,000.00 | 30,000 |
| Bio-Plex assays | 22,000 | 11,000 | 33,000 |
| In vitro activation assays | 15,000 | 7,500 | 22,500 |
| ELISA kits (sCD14: \$700, sCD163: \$900, neopterin: β-microglobulin: \$910; chitotriosidase: \$600): \$2,510 | 3,110 | 1,555 | 4,665 |
| Other Supplies | | | |
| Center For Clinical Trials fee | 1,000 | | 1,000 |
| Patient reimbursement | 2,400 | 600 | 3,000 |
| Personnel (3% COLA for year 2) | | | |
| PI (W. Royal; 5% effort) | 15,000 | 15,450 | 30,450 |
| Co-Investigator (B. Stern; 1% effort) | 4,000 | 4,120 | 8,120 |
| Coordinator (15% effort) | 20,000 | 20,600 | 40,600 |
| Technical (15% effort) | 9,500 | 9,785 | 19,285 |
| Administrative (5%) | 3,500 | 3,605 | 7,105 |
| Total direct costs | 164,690 | 123,610 | 288,300 |
| Indirect costs (30%) | 47,703 | 34,865 | 82,568 |
| IRB fee | 2,000 | 1,000 | 3,000 |
| TOTAL | 212,393 | 158,475 | 370,868 |

Please submit your curriculum vitae with the investigator initiated concept to your MSL and/or email to <a href="mailto:studyinfo@questcor.com">studyinfo@questcor.com</a>.



#### 11. References

- Agostini, C, Meneghin, A, Semenzato, G (2002). T-lymphocytes and cytokines in sarcoidosis. Curr. Opin. Pulm. Med., 8, 435-440.
- Arnason, BG, Berkovich, R, Catania, A, Lisak, RP, Zaidi, M (2013). Mechanisms of action of adrenocorticotropic hormone and other melanocortins relevant to the clinical management of patients with multiple sclerosis. Mult. Scler., 19, 130-136.
- Co, DO, Hogan, LH, Il-Kim, S, Sandor, M (2004). T cell contributions to the different phases of granuloma formation. Immunol. Lett., 92, 135-142.
- Judson, MA, Costabel, U, Drent, M, Wells, A, Maier, L, Koth, L, Shigemitsu, H, Culver, DA, Gelfand, J, Valeyre, D, Sweiss, N, Crouser, E, Morgenthau, AS, Lower, EE, Azuma, A, Ishihara, M, Morimoto, S, Tetsuo, YT, Shijubo, N, Grutters, JC, Rosenbach, M, Li, HP, Rottoli, P, Inoue, Y, Prasse, A, Baughman, RP, Organ Assessment Instrument Investigators TW (2014). The WASOG Sarcoidosis Organ Assessment Instrument: An update of a previous clinical tool. Sarcoidosis. Vasc. Diffuse. Lung Dis., 31, 19-27.
- Miller, DH, Kendall, BE, Barter, S, Johnson, G, MacManus, DG, Logsdail, SJ, Ormerod, IE, McDonald, WI (1988). Magnetic resonance imaging in central nervous system sarcoidosis. Neurology, 38, 378-383.
- Miyara, M, Amoura, Z, Parizot, C, Badoual, C, Dorgham, K, Trad, S, Kambouchner, M, Valeyre, D, Chapelon-Abric, C, Debre, P, Piette, JC, Gorochov, G (2006). The immune paradox of sarcoidosis and regulatory T cells. J. Exp. Med., 203, 359-370.
- Moller, DR (2003). Treatment of sarcoidosis -- from a basic science point of view. J. Intern. Med., 253, 31-40.
- Royal, W, III, Mia, Y, Li, H, Naunton, K (2009). Peripheral blood regulatory T cell measurements correlate with serum vitamin D levels in patients with multiple sclerosis. J. Neuroimmunol., 213, 135-141.
- Royal, W, III, Wang, H, Jones, O, Tran, H, Bryant, JL (2007). A vitamin A deficient diet enhances proinflammatory cytokine, Mu opioid receptor, and HIV-1 expression in the HIV-1 transgenic rat. J. Neuroimmunol., 185, 29-36.
- Royal, W, III, Zhang, L, Guo, M, Jones, O, Davis, H, Bryant, JL (2012). Immune activation, viral gene product expression and neurotoxicity in the HIV-1 transgenic rat. J Neuroimmunol., 247, 16-24.
- Shi, C, Pamer, EG (2011). Monocyte recruitment during infection and inflammation. Nat. Rev. Immunol., 11, 762-774.
- Stern, BJ, Aksamit, A, Clifford, D, Scott, TF (2010). Neurologic presentations of sarcoidosis. Neurol. Clin., 28, 185-198.
- Stern, BJ, Krumholz, A, Johns, C, Scott, P, Nissim, J (1985). Sarcoidosis and its neurological manifestations. Arch. Neurol., 42, 909-917.

